CLINICAL TRIAL: NCT07032012
Title: The Impact of Pre-anesthetic Evaluation on the Anxiety of Orthopedic Patients: a Randomized Clinical Trial.
Brief Title: Impact of Pre-anesthetic Evaluation on the Anxiety
Acronym: iPAEonAnx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, TSA, MSc, PhD, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: iPAEonAnx
Record Dates: First submitted 2025-04-30; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Postoperative Care; Preoperative Anxiety
Keywords: Anesthesia; Orthopedics; Anxiety; Postoperative
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control - anxiety evaluation before Pre-anesthetic (Other): If allocated to the group control, the anxiety questionnaire will be applied, and then the pre-anesthetic evaluation will be conducted.
  Interventions: Other: control - anxiety evaluation before Pre-anesthetic; Other: group intervention - anxiety evaluation after Pre-anesthetic
- intervention - anxiety evaluation after Pre-anesthetic (Active Comparator): If allocated to the group intervention, the first contact of the participant with the interviewer will be on the eve of surgery, in the ward. At that moment, the pre-anesthetic evaluation will be conducted. The next day, upon admission to the preoperative room, the anxiety questionnaire will be applied.
  Interventions: Other: control - anxiety evaluation before Pre-anesthetic; Other: group intervention - anxiety evaluation after Pre-anesthetic

INTERVENTIONS:
Other: control - anxiety evaluation before Pre-anesthetic — If allocated to the group control, the anxiety questionnaire will be applied, and then the pre-anesthetic evaluation will be conducted.
Other: group intervention - anxiety evaluation after Pre-anesthetic — If allocated to the group intervention, the first contact of the participant with the interviewer will be on the eve of surgery, in the ward. At that moment, the pre-anesthetic evaluation will be conducted. The next day, upon admission to the preoperative room, the anxiety questionnaire will be applied.

SUMMARY:
Since the last century, it has been understood that "the pre-anesthetic evaluation is the patient's right and the anesthesiologist's duty." As early as 2006, the Conselho Federal de Medicina (CFM) published a resolution addressing the anesthetic act and guiding the conduct of pre-anesthetic evaluation (PAE) and in 2017 revised these guidelines in a new resolution. The PAE is an important step in preparing the patient for elective surgical procedures. It refers to the moment when the anesthesiologist and patient have the opportunity to get to know each other, optimize the patient's clinical conditions and even request exams or consult other specialists when necessary. The prevalence and levels of anxiety, commonly generated by the expectation of the surgical-anesthetic procedure, tend to reduce with the PAE. This leads to fewer patients presenting to the operating room with arterial hypertension or arrhythmia, which are triggered by anxiety. It can be said that the implementation of the PAE directs screening processes and consequently reduces the patient's risk to unnecessary procedures or consultations. It also highlights the reduction in perioperative morbidity and mortality rates. By analyzing the dynamics of the surgical center, where the space is highly technological and contested by various surgical specialties, it is possible to associate the PAE with the reduction in cancellation rates of procedures and the proper use of space. Measuring sentiment is difficult and to assess anxiety, one can use complex questionnaires to small and objective scales. Some studies show how anxiety can contribute to increased postoperative pain, higher medication consumption, and longer hospitalization time. A possible tool to change this scenario would be the PAE, but its relationship with anxiety still needs to be further documented, especially in Brazil. Therefore, this project seeks to study the hypothesis that the PAE reduces anxiety levels, brings quality to the anesthetic-surgical experience, and improves perioperative morbidity indicators. This study aims to evaluate the impact of pre-anesthetic evaluation on perioperative surgical outcomes in patients of the orthopedic specialty undergoing procedures at the institution. It aims to identify the anxiety level of patients undergoing orthopedic surgery. This randomized clinical trial will be conducted at the Hospital de Base do Distrito Federal, Brasília, Distrito Federal, Brazil.

ELIGIBILITY:
Inclusion Criteria:

* elective or urgent orthopedic surgery
* aged between 18 and 65 years
* ASA classification I to III

Exclusion Criteria:

* Patient refusal to participate
* Patient refusal to sign the IC
* Lack of education
* History of psychiatric illness, especially depression
* Limited cognitive capacity (self-declared or informed by a companion)
* Prolonged hospitalization (greater than or equal to 14 days)
* Emergency surgery
* Inability to understand the IC.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pre operative anxiety levels | Before the procedure.
  Assessment of pre operative anxiety levels using the State-Trait Anxiety Inventory - anxiety scale in patients who will or will not receive pre-anesthesia assessment in orthopedic surgeries. The score on this scale ranges from 10 to 40, with 10 being the calmest possible individual and 40 being the most anxious possible.

SECONDARY OUTCOMES:
Assess anxiety levels using the Likert scale | Before the procedure
  Assess anxiety levels using the Likert scale. This scale has a drawing of 5 faces that range from very anxious (on the left) to very calm (on the right)

REFERENCES:
- [Background] Ambulkar R, Patel A, Patil S, Savarkar S. Patient satisfaction with anaesthesia services in a tertiary care cancer centre. (SAY study). J Anaesthesiol Clin Pharmacol. 2022 Jan-Mar;38(1):111-117. doi: 10.4103/joacp.JOACP_187_20. Epub 2022 Jan 12. PMID 35706652